CLINICAL TRIAL: NCT01222286
Title: Multicenter Phase II Study on the Anti-tumor Activity, Safety and Pharmacology of Two Dose Regimens of IPH2101, a Fully Human Monoclonal Anti KIR Antibody, in Patients With Smoldering Multiple Myeloma (KIRMONO)
Brief Title: Study on the Anti-tumor Activity, Safety and Pharmacology of IPH2101 in Patients With Smoldering Multiple Myeloma
Acronym: KIRMONO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPH2101-203; NCT01960959 (obsolete NCT alias)
Record Dates: First submitted 2010-10-08; First posted 2010-10-18 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Smoldering Multiple Myeloma
Keywords: Smoldering Multiple Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — IPH-2101

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPH2101 0.2 mg/kg (Experimental): 0.2 mg/Kg every 4 weeks by intravenous route over 1 hour, for 6 or up to 12 cycles
  Interventions: Drug: IPH2101
- IPH2101 2 mg/kg (Experimental): 2 mg/Kg every 4 weeks by intravenous route over 1 hour, for 6 or up to 12 cycles
  Interventions: Drug: IPH2101

INTERVENTIONS:
Drug: IPH2101 — 0.2 mg/Kg or 2mg/Kg, every 4 weeks by intravenous route over 1 hour, for 6 or up to 12 cycles
  Other Names: a human monoclonal anti-KIR antibody (1-7F9)

SUMMARY:
The purpose of this study is to evaluate the anti-tumor activity, safety and pharmacology of two dose regimens (0.2 and 2 mg/kg)of IPH2101 in patients with Smoldering Multiple Myeloma.

DETAILED DESCRIPTION:
This is a randomized Phase II, open label, multi-centre study, with two independent arms.

Patients receive 6 injections of IPH2101, at the dose of 0.2 mg/kg or 2 mg/kg (according to their randomization) administered over one hour infusion at four weeks intervals.

A patient whose disease achieves at least a minimal response to study treatment at any time during the initial period of 6 cycles can be treated with an additional period of treatment of 6 cycles.

Patients are followed 6 months after treatment completion or until a KIR occupancy level < 30% (i.e if the time required for KIR desaturation was > 6 months), whichever is longer.

ELIGIBILITY:
Inclusion Criteria:

1. SMM of any risk level according to a definition derived of the International Myeloma Working Group definition ( Br J Haematol 2003; 121: 749) : Serum M protein ≥ 3 g/dl , AND/OR Bone Marrow plasma cells ≥ 10 % with no evidence of end-organ damage (CRAB)

   * (C)Absence of hypercalcemia : Ca < 10.5 mg/dl
   * (R)Absence of renal failure : creatinine < 2mg/dl (177 μmol/l) or calculated creatinine clearance(according to MDRD) > 50 ml/min
   * (A)Absence of anemia : Hb > 11 g/dl
   * (B)Absence of lytic bone lesion on standard skeletal survey (MRI could be used if clinically indicated)
2. Measurable disease defined as a disease with a serum M protein ≥ 1 g/dl
3. No evidence of fatigue, recurrent infections or any clinical suspicion of MM
4. Diagnosis of SMM confirmed on two consecutive assessments (ie fluctuation under 25% of serum protein level) performed with at least a 4 week interval.
5. Age > 18 years or < 75 years
6. ECOG performance status of 0 or 1
7. Male or female patient who accepts and is able to use recognised effective contraception (oral contraceptives, IUCD, barrier method of contraception in conjunction with spermicidal jelly) throughout the study when relevant
8. Informed consent signed by the patient

Exclusion Criteria:

1. Previous treatment having a proven or potential impact on myelomatous cells proliferation or survival (including IMiDs or proteasome inhibitors, conventional chemotherapies within the last 5 years, steroids within the last month prior to enrolment). Previous bisphosphonates started less than 3 months prior to enrolment.
2. Use of any investigational agent within the last 3 months
3. Clinical laboratory values at screening

   * Platelet < 75 x 10^9 /l
   * ANC < 1.5 x 10^9 /l
   * Bilirubin levels >1.5 ULN ; ALT and AST > 3 ULN (grade 1 NCI)
4. Primary or associated amyloidosis
5. Abnormal cardiac status with any of the following

   1. NYHA stage III or IV congestive heart failure
   2. myocardial infarction within the previous 6 months
   3. symptomatic cardiac arrhythmia requiring treatment or persisting despite appropriate treatment
6. Current active infectious disease or positive serology for HIV, HCV or positive Hbs Antigen
7. History of or current auto-immune disease
8. History of other active malignancy within the past five years (apart from basal cell carcinoma of the skin, or in situ cervix carcinoma).
9. Serious concurrent uncontrolled medical disorder
10. History of allograft or solid organ transplantation
11. Pregnant or lactating women
12. Any condition potentially hampering compliance with the study protocol and follow-up schedule

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Munshi, MD, Principal Investigator — Dana-Farber Cancer Institute- Medical Oncology- Boston MA-USA
Locations (5):
- United States (5):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mount Sinai School of Medicine, New York, New York
  - Ohio State University, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 44 patients screened, 14 subjects were not randomized, 12 of whom were screen failures, 30 patients randomized.
Pre-assignment Details: All patients enrolled were screened in order to verify the inclusion/exclusion criteria. All patients enrolled (30 patients) were analyzed.
Period: Overall Study
Arm/Group | IPH2101 0.2 mg/kg | IPH2101 2 mg/kg
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IPH2101 0.2 mg/kg | IPH2101 2 mg/kg | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (7.62) | 58.4 (13.11) | 61.2 (10.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 7 | 10 | 17
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Rate of Patients Achieving an Objective Response
Description: The primary end point is the rate of patients achieving an objective response (defined according to the International Myeloma Working Group uniform response criteria), including minimal response, (as derived from the European Society for Blood and Marrow Transplantation criteria), achieved at any time until end of study and confirmed on two consecutive assessments at 4 weeks interval.
Time Frame: from start to end of study (14 months)
Population: The ITT population included all randomized subjects.
Measure: Number; unit: participants
Arm/Group | IPH2101 0.2 mg/kg | IPH2101 2 mg/kg
Number analyzed (Participants) | 16 | 14
participants | 0 | 0

2. Secondary Outcome: Safety Assessment
Description: adverse events, physical examination and biological changes during the whole clinical trial.
Time Frame: Adverse events collected from screening visit (date of signature of Inform Consent Form) up to the End of Study, up to 14 months
Population: The safety population included all subjects who received at least 1 dose of IPH2101
Measure: Number; unit: Patients with any AE
Arm/Group | IPH2101 0.2 mg/kg | IPH2101 2 mg/kg
Number analyzed (Participants) | 16 | 14
Patients with any AE | 16 | 14

3. Secondary Outcome: Pharmacodynamics of IPH2101
Description: biological activity of IPH2101 on KIR occupancy at End of Treatment
Time Frame: from start to end of study (14 months)
Population: all subjects who received at least 1 dose of IPH2101
Measure: Mean (Full Range); unit: % of occupancy of killer like receptor
Arm/Group | IPH2101 0.2 mg/kg | IPH2101 2 mg/kg
Number analyzed (Participants) | 9 | 11
% of occupancy of killer like receptor | 73.1 [46 to 98] | 92 [80 to 96]

4. Secondary Outcome: Secondary Anti-tumor Activity
Description: * any change of M-protein in serum occurring during the study (>25 percentage increase in level of serum M-protein)
  * progression to active Multiple Myeloma
  Definition of active Multiple Myeloma: Evidence of progression based on the IMWG criteria for progressive disease in myeloma and any one or more of the following felt related to the underlying clonal plasma cell proliferative disorder :
  * Development of new soft tissue plasmacytomas or bone lesions
  * Hypercalcemia (> 11mg/100ml)
  * Decrease in hemoglobin of > 2g/100ml
  * Rise in serum creatinine by 2 mg/100ml or more
Time Frame: from start to end of study (14 months)
Measure: Number; unit: Participant
Arm/Group | IPH2101 0.2 mg/kg | IPH2101 2 mg/kg
Number analyzed (Participants) | 16 | 14
Participant
  serum M-protein progression | 4 | 8
  Progression to active Multiple Myeloma | 2 | 3

ADVERSE EVENTS:
Time Frame: Adverse events related to Study Drug, collected from screening visit (date of signature of Inform Consent Form) up to the End of Study, up to 14 months
Arm/Group | IPH2101 0.2 mg/kg | IPH2101 2 mg/kg
Serious Adverse Events (participants affected / at risk) | 2/16 | 0/14
Other Adverse Events (participants affected / at risk) | 12/16 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IPH2101 0.2 mg/kg (N=16) | IPH2101 2 mg/kg (N=14)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) — This event was assessed as possibly related to study treatment
Demyelinating polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) — This event was assessed as unlikely related to study treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IPH2101 0.2 mg/kg (N=16) | IPH2101 2 mg/kg (N=14)
Fatigue (General disorders) | 5 (5) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Chills (General disorders) | 2 (2) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Edema Peripheral (General disorders) | 0 (0) | 2 (2)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
neutrophil count decreased (Investigations) | 1 (1) | 2 (2)
blood creatinine increased (Investigations) | 2 (2) | 0 (0)
white blood cell count decreased (Investigations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
seasonal allergy (Immune system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No